CLINICAL TRIAL: NCT03031041
Title: Comparison of Difference Hydrodissection Technique in Patients With Carpal Tunnel Syndrome
Brief Title: Comparison of Difference Hydrodissection for CTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Yung-Tsan Wu, Attending Physician of Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Difference PIT for CTS
Record Dates: First submitted 2017-01-21; First posted 2017-01-25 (Estimated); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Hydrodissection; short-axis; long-axis
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short-axis hydrodissection (Experimental): Ultrasound-guided short-axis hydrodissection with normal saline between carpal tunnel and median nerve
  Interventions: Procedure: Ultrasound-guided short-axis hydrodissection with 5cc normal saline
- Long-axis hydrodissection (Active Comparator): Ultrasound-guided long-axis hydrodissection with normal saline between carpal tunnel and median nerve
  Interventions: Procedure: Ultrasound-guided long-axis hydrodissection with 3cc normal saline

INTERVENTIONS:
Procedure: Ultrasound-guided short-axis hydrodissection with 5cc normal saline — Ultrasound-guided short-axis hydrodissection with 5cc normal saline between carpal tunnel and median nerve
  Arms: Short-axis hydrodissection
Procedure: Ultrasound-guided long-axis hydrodissection with 3cc normal saline — Ultrasound-guided long-axis hydrodissection with 3cc normal saline between carpal tunnel and median nerve
  Arms: Long-axis hydrodissection

SUMMARY:
Carpal tunnel syndrome (CTS) is the most common peripheral entrapment neuropathy with involving compression of the median nerve in the carpal tunnel. Rather than other progressive disease, CTS is characterized by remission and recurrence. The hydrodissection could decrease the entrapment of nerve to restore blood supply. Despite the hydrodissection was pervasively used in clinical practice, current researches contain small participant without control group or randomized leading to foreseeable selection bias. The investigators design a randomized, double-blind, controlled trial to assess the effect of different method of ultrasound-guided hydrodissection in patients with CTS.

DETAILED DESCRIPTION:
After obtaining written informed consent, patients with bilateral CTS will been randomized into intervention and control group. Participants in short-axis group received one-dose ultrasound-guided hydrodissection with short-axis approach and long-axis group received one-dose ultrasound-guided injection with long-axis approach. No additional treatment after injection through the study period. The primary outcome is Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) and secondary outcomes include visual analog scale (VAS), cross-sectional area (CSA) of the median nerve, sensory nerve conduction velocity of the median nerve, and finger pinch strength. The evaluation was performed pretreatment as well as on the 2nd week, 1st, 2nd, 3rd and 6th month after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-80 year-old.
* Diagnosis was confirmed using an electrophysiological study

Exclusion Criteria:

* Cancer
* Coagulopathy
* Pregnancy
* Inflammation status
* Cervical radiculopathy
* Polyneuropathy, brachial plexopathy
* Thoracic outlet syndrome
* Previously undergone wrist surgery or steroid injection for CTS

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline of severity of symptoms and functional status on 2nd week, 1st, 2nd, 3rd and 6th month after injection | Pre-treatment, 2nd week, 1st, 2nd, 3rd and 6th month after injection
  Boston carpal tunnel syndrome questionnaire (BCTQ) is a frequently used patient-based questionnaire for measurement of CTS which encompasses two components. In total, 11 questions and 8 items were evaluated to rate the symptom severity scale (SSS) and functional status scale (FSS), respectively. Both subscales range from 1 to 5 with a higher score indicating a higher degree of disability. The mean of total SSS and FSS divided with each item score were used for further analysis.

SECONDARY OUTCOMES:
Change from baseline of pain on 2nd week, 1st, 2nd, 3rd and 6th month after injection | Pre-treatment, 2nd week, 1st, 2nd, 3rd and 6th month after injection
  Digital pain severity or paresthesia/dysthesia was evaluated using visual analog scale (VAS). Pain score scale ranged from 0 to 10, with 10 indicating the most severe pain.
Change from baseline of cross-sectional area of the median nerve on 2nd week, 1st, 2nd, 3rd and 6th month after injection | Pre-treatment, 2nd week, 1st, 2nd, 3rd and 6th month after injection
  Using the musculoskeletal sonogram to measure the cross-sectional area of the median nerve before treatment and multiple time frame after treatment.
Change from baseline of conduction velocity, amplitude of median nerve on 2nd week, 1st, 2nd, 3rd and 6th month after injection | Pre-treatment, 2nd week, 1st, 2nd, 3rd and 6th month after injection
  Electrophysiological study of the median nerve before treatment and multiple time frame after treatment.
Change from baseline of finger pinch on 2nd week, 1st, 2nd, 3rd and 6th month after injection | Pre-treatment, 2nd week, 1st, 2nd, 3rd and 6th month after injection
  The finger pinch strength was measured using dynamometer (Fabrication Enterprises Inc., USA). The subject was seated with shoulder adducted and neutrally rotated with the elbow flexed at 90°. The forearm and wrist were positioned in a neutral position for the palmar pinch

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Tsan Wu, MD, Principal Investigator — Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital
Locations (1):
- Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital, Taipei, Neihu District, Taiwan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] DeLea SL, Chavez-Chiang NR, Poole JL, Norton HE, Sibbitt WL Jr, Bankhurst AD. Sonographically guided hydrodissection and corticosteroid injection for scleroderma hand. Clin Rheumatol. 2011 Jun;30(6):805-13. doi: 10.1007/s10067-010-1653-6. Epub 2011 Jan 15. PMID 21234632
- [Background] Mulvaney SW. Ultrasound-guided percutaneous neuroplasty of the lateral femoral cutaneous nerve for the treatment of meralgia paresthetica: a case report and description of a new ultrasound-guided technique. Curr Sports Med Rep. 2011 Mar-Apr;10(2):99-104. doi: 10.1249/JSR.0b013e3182110096. PMID 21623291
- [Result] Smith J, Wisniewski SJ, Finnoff JT, Payne JM. Sonographically guided carpal tunnel injections: the ulnar approach. J Ultrasound Med. 2008 Oct;27(10):1485-90. doi: 10.7863/jum.2008.27.10.1485. PMID 18809959
- [Result] Cass SP. Ultrasound-Guided Nerve Hydrodissection: What is it? A Review of the Literature. Curr Sports Med Rep. 2016 Jan-Feb;15(1):20-2. doi: 10.1249/JSR.0000000000000226. PMID 26745165